CLINICAL TRIAL: NCT04972032
Title: Prevention of Postoperative Adhesion Recurrence by Estrogen-intrauterine Stent System
Brief Title: Efficacy of Estrogen-intrauterine Stent System After Intrauterine Adhesiolysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Limin Feng (Other)
Responsible Party: Sponsor-Investigator, Limin Feng, director, Beijing Tiantan Hospital
Organization: Beijing Tiantan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-IUS
Record Dates: First submitted 2021-06-30; First posted 2021-07-22 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Intrauterine Adhesion
Keywords: Intrauterine adhesion; recurrence; estrogen; intrauterine stent
MeSH Terms: conditions — Gynatresia; Recurrence

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Estrogen Intrauterine Stent System (Experimental): An Intrauterine Stent System with estrogen will be introduced into the uterine cavity after TCRA(transcervical resection of adheison).
  Interventions: Device: Estrogen Intrauterine Stent System
- Foley balloon combined with self-cross-link sodium hyaluronate gel (Other): Subjects will be given Foley balloon (manufacturer: Zhanjiang Star Enterprise Co., Ltd.) combined with self-cross-linked sodium hyaluronate gel (manufacturer: BioRegen Biomedical (Changzhou) Co., Ltd.) after TCRA surgery.
  Interventions: Device: Foley balloon combined with self-cross-link sodium hyaluronate gel

INTERVENTIONS:
Device: Estrogen Intrauterine Stent System — A Estrogen Intrauterine Stent System（E-IUS）will be introduced post-operatively. The E-IUS will be removed 60 days after surgery with continuous dydrogesterone administration for 5 days at 20 mg/d, and routine management.
  Arms: Estrogen Intrauterine Stent System
Device: Foley balloon combined with self-cross-link sodium hyaluronate gel — Foley balloon combined with self-crosslinking sodium hyaluronate gel will be introduced post-operatively，2 cycles of estrogen-progestin sequential therapy comprised of continuous estrogen and progestin added in the second half of the cycle or continuous estradiol valerate for 60 days, followed by dydrogesterone for 10 days
  Arms: Foley balloon combined with self-cross-link sodium hyaluronate gel

SUMMARY:
This is a prospective, randomized, single-blinded,multi-center trial to compare the efficacy of an Estrogen-intrauterine stent system with foley balloon combined with intrauterine cross-linked sodium hyaluronate gel in the prevention of intrauterine adhsion recurrence after hysteroscopic adhesiolysis.

DETAILED DESCRIPTION:
Patients suspect to be suffering from IUA will be recruited following a systematic pre-operative assessment process. This will include a detailed history of the menstrual pattern, previous intrauterine surgery, and reproductive history, as well as 3D transvaginal ultrasound. The severity and extent of intrauterine adhesions will be scored according to the AFS score. All patients will receive hysteroscopic adhesiolysis with the aid of ultrasound guidance as necessary. After adhesiolyis, the patients will assigned to two groups randomly,namely,the E-IUS(estrogen intrauterine stent system) group and the control group. Adhesion will be evaluated by hysteroscopy at second-look hysteroscopy before 60 after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 18-40 years;

  * Meets the diagnostic criteria for moderate to severe uterine adhesions;

    * Has the indication for TCRA surgery and is intending to undergo TCRA surgery;

      * Female subjects are not breastfeeding at the time of the screening visit; ⑤ Voluntary acceptance of the treatment and has signed the informed consent form.

Exclusion Criteria:

* Known allergic reactions to or contraindications for silicone rubber materials, estradiol and its metabolites, Foley balloon catheters and/or intrauterine cross-linked sodium hyaluronate gel;

  * Presence of contraindications for TCRA surgery;

    * Requires oral hormonal medications for a prolonged period of time;

      * Has used high-dose estrogen medication within one month prior to surgery;

        * Suffering from diseases such as genital tract tuberculosis, acute genital tract inflammation, pelvic inflammatory disease, abnormal uterine bleeding caused by systemic disease or malignant tumours of the genital organs; ⑥ Perimenopausal and menopausal females;

          ⑦ Comorbid with severe primary diseases of the cardiovascular, cerebrovascular, hepatic, renal or hematopoietic system, or peptic ulcer disease, or severe diseases affecting patient survival (such as tumours or AIDS), or mental illness;

          ⑧ Drug or alcohol dependence;

          ⑨ Has enrolled in other clinical trials within the last 1 month;

          ⑩ Patients with factors considered by the investigators to be unsuitable for enrollment.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — The female patients after TCRA surgery
Enrollment: 246 (Estimated)
Dates: Start 2020-09-02 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Post-operative adhesion recurrence rate(%) | 60 days
  The severity of adhesion will be assessed by hysteroscopy before and on d60 after surgery using the America Fertility Score (AFS) system. If the AFS score on D60 second-look hysteroscopy over 0 will be considered as adhesion recurrence. Post-operative adhesion recurrence rate(%)=(patients whose AFS score >0-point after surgery/All patients after surgery)X100%. The recurrence rate (%) is range from 0(Mini) to 100(Max).The lower the recurrence means the patient has a better post-operative outcome.

SECONDARY OUTCOMES:
Menstrual improvement rate %(PBAC score) | 60 days
  Menstrual improvement rate (evaluated by PBAC score) on 60 days after surgery
Pregnancy rate% | 1-2 years
  Pregnancy rate%=Number of patients with successful Pregnancy /Number of all patients）X100%

CONTACTS AND LOCATIONS:
Overall Officials: Limin Feng, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- YiPuRun (Shanghai) Biotechnology Co.,Ltd., Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Feng L, Sun Y, Zhang S, Qian Y, Fang S, Yang B, Xu L, Li J, Niu Y, Zhang S, Zhang L, Chen J. A novel intrauterine estrogen-releasing system for preventing the postoperative recurrence of intrauterine adhesion: a multicenter randomized controlled study. BMC Med. 2024 Sep 16;22(1):395. doi: 10.1186/s12916-024-03608-4. PMID 39285313